CLINICAL TRIAL: NCT03797599
Title: The Effects of Length of Mindfulness Practice on Mindfulness, Depression, Anxiety and Stress: A Randomised Controlled Experiment
Brief Title: Study Examining the Effects of Mindfulness and Similar Audio-guided Exercises.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S_Strohmaier_29-11-18
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-09

CONDITIONS: Mindfulness; Healthy Population

STUDY DESIGN:
Masking Description: Participants will be masked to the extent that they will not be told which group they have been allocated to nor the exact nature of the the three groups. However, they will be aware of the exercises they are asked to undertake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 minutes of mindfulness practice (Experimental): Two sessions a week for two weeks of: 5 minutes listening to audio book excerpts followed by 20 minutes of audio guided mindfulness practice. Participants will be asked not to engage in formal mindfulness practice outside of these sessions during the study.
  Interventions: Behavioral: 20 minutes of mindfulness practice; Other: 5 minute audio book
- 5 minutes of mindfulness practice (Active Comparator): Two sessions a week for two weeks of: 20 minutes listening to audio book excerpts followed by 5 minutes of audio guided mindfulness practice. Participants will be asked not to engage in formal mindfulness practice outside of these sessions during the study.
  Interventions: Behavioral: 5 minutes of mindfulness practice; Other: 20 minute audio book
- Audio book control (Placebo Comparator): Two sessions a week for two weeks of: 25 minutes listening to audio book excerpts (with non mindfulness practice). Participants will be asked not to engage in formal mindfulness practice during the study.
  Interventions: Other: 25 minute audio book

INTERVENTIONS:
Behavioral: 20 minutes of mindfulness practice — A 20 minute audio guided mindfulness of breathing practice per session, for four sessions.
  Arms: 20 minutes of mindfulness practice
Behavioral: 5 minutes of mindfulness practice — A 5 minute audio guided mindfulness of breathing practice per session, for four sessions.
  Arms: 5 minutes of mindfulness practice
Other: 5 minute audio book — 5 minutes from an audio book by Bill Bryson ('A Short History of Nearly Everything') per session, for four sessions.
  Arms: 20 minutes of mindfulness practice
Other: 20 minute audio book — 20 minutes from an audio book by Bill Bryson ('A Short History of Nearly Everything'), per session, for four sessions.
  Arms: 5 minutes of mindfulness practice
Other: 25 minute audio book — 25 minutes from an audio book by Bill Bryson ('A Short History of Nearly Everything'), per session, for four sessions.
  Arms: Audio book control

SUMMARY:
This study aims to examine whether greater length of mindfulness practice results in more beneficial outcomes.

DETAILED DESCRIPTION:
This study will randomise participants to one of three groups: (1) four sessions of medium length mindfulness practice (lasting 20 mins) and 5 mins of an audio book; (2) four sessions of brief mindfulness practice (lasting 5 mins) and 20 mins of an audio book; and (3) a control group who just receive 4 sessions of audio book (lasting 25 mins). In the mindfulness arms, in each session, the participants will receive the audio book prior to the mindfulness practice. Mindfulness levels, and depression, anxiety and stress will be measured by self-report at baseline, session by session, and at post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Members of the general public, especially university students or staff.
* Adequate understanding of spoken and written English

Exclusion Criteria:

* Currently experiencing significant difficulties with their mental wellbeing.
* Currently have a personal mindfulness practice.
* Currently participating in a mindfulness-based intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline at post-intervention (week 3) on the Five Factor Mindfulness Questionnaire -15 item version (FFMQ-15) | Post-intervention (3 weeks after baseline).
  The Five Factor Mindfulness Questionnaire -15 item version is a self-report measure of mindfulness, producing a total score between 15 and 75, with higher scores indicating greater levels of mindfulness. (Note that the observe subscale will be excluded from the calculation of the total score, as recommended in https://doi.org/10.1002/jclp.21865 and http://dx.doi.org/10.1037/pas0000263 producing a total score between 12 and 60).

SECONDARY OUTCOMES:
Change from baseline at post-intervention (week 3) on the Depression, Anxiety and Stress Scale - 21 item version (DASS-21). | Post-intervention (3 weeks after baseline).
  The Depression, Anxiety and Stress Scale - 21 is a self-report measure of depression, anxiety and stress, producing a total score between 0 and 63, with higher scores indicating greater symptomatology.

OTHER OUTCOMES:
Sessional Five Factor Mindfulness Questionnaire -15 item version (FFMQ-15) scores. | Baseline, session 2 (week 1), session 3 and 4 (week 2), and post-intervention (week 3).
  The FFMQ-15 (described above) will be administered at the start of the first session (baseline), immediately after sessions 2 (week 1), 3 (week 2) and 4 (week 2), and at post-intervention (week 3), to examine patterns in changes in mindfulness over the course of the study.
Sessional Depression, Anxiety and Stress Scale - 21 item version (DASS-21) scores | Baseline, session 2 (week 1), session 3 and 4 (week 2), and post-intervention (week 3).
  The DASS-21 (described above) will be administered at the start of the first session (baseline), immediately after sessions 2 (week 1), 3 (week 2) and 4 (week 2), and at post-intervention (week 3), to to examine patterns in changes over the course of the study.
Session 1 Toronto Mindfulness Scale (TMS). | Session 1 (week 1).
  The TMS is a 13-item self-report measure of state mindfulness that produces scores for curiosity and decentering. The curiosity score ranges from 0 to 24, the decentering score from 0 to 28, and the total score from 0 to 52, with higher scores indicating greater curiosity, decentering and overall state mindfulness respectively.
Session 2 Toronto Mindfulness Scale (TMS). | Session 2 (week 1).
  As described above.
Session 3 Toronto Mindfulness Scale (TMS). | Session 3 (week 2).
  As described above.
Session 4 Toronto Mindfulness Scale (TMS). | Session 4 (week 2).
  As described above.

CONTACTS AND LOCATIONS:
Overall Officials: Fergal Jones, PhD, PsychD, Study Director — Canterbury Christ Church University; James Cane, PhD, Study Director — Canterbury Christ Church University; Sarah Strohmaier, MSc, Principal Investigator — Canterbury Christ Church University
Locations (1):
- Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided